CLINICAL TRIAL: NCT02088242
Title: Physiological and Molecular Influences of Astaxanthin Supplementation on Heat Strain in Humans
Acronym: Astaxanthin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofir Frenkel MD, head investigator of Heller institute of physiology, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SHEBA-13-0471-BA-CTIL; IDF-1295-2013 (Other: IDF)
Record Dates: First submitted 2014-03-03; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Body Temperature Regulation
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects receiving placebo will be asked to ingest 3 capsules identical in shape, colour and size to the Astaxanthin capsules, and will contain only the inactive ingredients of the same formulation.
  Interventions: Drug: Placebo
- Astaxanthin (Experimental): Subjects receiving Astaxanthin will be asked to ingest 3 capsules containing 4mg of Astaxanthin each (a daily dose of 12mg).
  Interventions: Drug: Astaxanthin

INTERVENTIONS:
Drug: Astaxanthin — Oral supplementation with the food supplement Astaxanthin. Subjects receiving Astaxanthin will be asked to ingest 3 capsules containing 4mg of Astaxanthin each (a daily dose of 12mg).
  Arms: Astaxanthin
Drug: Placebo — 3 capsules identical in shape, colour and size to the Astaxanthin capsules, which contain only the inactive ingredients of the same formulation.
  Arms: Placebo

SUMMARY:
Exposure to heat stress can compromise the physiological and cognitive function and be life threatening, particularly in a military setting. Various strategies of precondition to heat stress that have been explored in the past proved to be inapplicable. We aim to examine the influences of Astaxanthin supplementation as a preconditioning strategy to heat stress in a human model using a heat tolerance test. This will be achieved by a double-blind, placebo controlled supplementation trial, exposing human subjects, before and after consuming Astaxanthin or a placebo, to a controlled heat strain environment, while performing moderate exercise in a heated chamber.

DETAILED DESCRIPTION:
34 young, healthy civilian volunteers will participate in this study. After reading and signing an informed consent form, all subjects will undergo medical examination and an interview with a nutritionist to assess their dietary intake of Astaxanthin. They will then undergo 3 days of training on the cognitive testing software.

During the first stage, while consuming an Astaxanthin free diet, the subjects will participate in the physiological tests:heat tolerance test (HTT), thermo-neutral test (TTT) and maximal oxygen consumption test (VO2max) on 3 separate days.

During the second stage, the subjects will be randomly and blindly assigned to either the placebo or the Astaxanthin supplementation arms, and undergo 35-40 days of supplementation.

Physiological testing of the second stage will take place between the 31st and 35th (up to 40th - optional) days of supplementation and will include HTT, TTT and VO2max on 3 separate days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy civilian volunteers.
* Aged 20-30 years.
* Without known medical illness or medication use.

Exclusion Criteria:

* The existence or suspicion of existing cardiac or respiratory disease.
* Hypertension.
* Diabetes.
* Any hormonal disease or any other chronic illness that may inhibit participation in the experiment.
* Infectious disease 3 days prior to the experiment.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Physiological strain | 2 months for each participant
  The physiological strain will be determined by monitoring body core temperature and heart rate of the subjects during a heat tolerance test (HTT) and a thermo-neutral test (TTT).The test is performed in a climatic chamber. During the test, the subject walks on a treadmill at a speed of 5 km/hr at a 2% grade for 2h. Body core temperature and heart rate are continuously monitored, and sweat rate is computed from body weight prior to and after the test, corrected for fluid intake.
Aerobic capacity | 2 months for each participant
  The aerobic capacity of the subjects will be determined by performing a maximal oxygen consumption test (VO2max). Volunteer's oxygen consumption (VO2) will be monitored continuously with a metabolic chart (ZAN- the name of the metabolic system), while running for 10 min on a treadmill under comfortable environmental conditions.

SECONDARY OUTCOMES:
Rectal temperature | 2 months for each participant
  The rectal temperature will be monitored by a rectal thermistor during each heat tolerance test (HTT) and thermo-neutral test (TTT) and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system (Biopac is the company in which the monitoring system was made).
Skin temperature | 2 months for each participant
  The skin temperature will be monitored by skin thermistors located at 3 sites (chest, arm and leg) and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.
Heart rate | 2 months for each participant
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).
Sweat rate | 2 months for each participant
  Sweat rate will be calculated from the patients' body weight and fluid balance.
Cognitive function | 2 months for each participant
  Cognitive function will be assessed using a cognitive testing software on laptop computers before and after performing the physiological tests.

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel-Hashomer, Ramat- Gan, Israel